CLINICAL TRIAL: NCT05679284
Title: The Prevalence and Predisposing Factors to Retained Drug Needle Fragments in People Who Inject Drugs: a Protocol for a Cross-sectional Observational Study
Brief Title: A Cross-Sectional Observational Study on Retained Drug Needle Fragments in People Who Use Intravenous Drugs
Status: Recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Deaconess Foundation (Unknown); A-Clinic Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: Retained drug needles
Record Dates: First submitted 2022-10-22; First posted 2023-01-10 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Drug Abuse, Intravenous; Substance Dependence; Needle Injury; Soft Tissue Injuries; Foreign Bodies
Keywords: Intravenous drug use; needle retention; needle fragment
MeSH Terms: conditions — Substance Abuse, Intravenous; Substance-Related Disorders; Soft Tissue Injuries; Foreign Bodies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Intravenous drug users with drug needle fragment retentions: All intravenous drug users from the service units will be asked to participate. X-ray imaging has the goal to identify patients with needle fragment retentions in subcutaneous tissue.
  Interventions: Radiation: Low-dose X-ray of subcutaneous tissues
- Controls: Intravenous drug users without drug needle fragment retentions: All intravenous drug users from the service units will be asked to participate. Control group consists of those with no radiologically confirmed subcutaneous needle fragment retentions.
  Interventions: Radiation: Low-dose X-ray of subcutaneous tissues

INTERVENTIONS:
Radiation: Low-dose X-ray of subcutaneous tissues — To identify needle fragment retentions, the radiologic imaging of all volunteers will be performed with X-ray using radiation doses as low as reasonably achievable (ALARA) and one projection per anatomic site.

SUMMARY:
In addition to the well-known toxicological harms of intravenous drug (IVD) use, there can also be local tissue complications, including infections, venous sclerosis, tissue necrosis, and drug needle fragment retentions. Drug needle fragments in subcutaneous tissue may cause local symptoms (usually pain and infections), but they have also been identified as causing emboli to organs. The literature has described numerous case reports of people who inject drugs (PWIDs) and have retained needle fragments. The prevalence of the condition is not known, and the researchers therefore aim to perform the first cross-sectional study of PWIDs to estimate how common needle fragment retentions are and what their risk factors are in this population.

DETAILED DESCRIPTION:
The clinical significance of retained needle fragments remains unknown. Needle retentions can be asymptomatic, cause local symptoms, and can sometimes even lead to dangerous complications such as needle emboli to the heart or lungs. The most common injection sites are likely the peripheral veins of the arms. However, continuous IVD use leads to vein sclerosis, and patients with long-term use may therefore also use peripheral veins of their lower limbs and even the central veins of the groin or neck. Subcutaneously retained needles can pose a risk of needlestick injury to medical staff during clinical examination and treatment procedures. Unrecognized retained needles can also cause hazards during magnetic resonance imaging.

The study protocol received a positive review from the Tampere University Hospital Ethics Committee (study code: R22037). The researchers subsequently received the organizational permissions necessary to conduct the study. PWIDs will be asked to give written informed consent prior to any study procedures. Participants will be asked to fill in a questionnaire about their basic information, drug use history, previous injection sites, and whether they have had any local complications due to injecting drugs. After the completion of the questionnaire, participants will undergo targeted X-ray imaging of the injection sites. As metallic objects, needle fragments can be visualized with standard X-ray imaging. Female participants of childbearing potential (< 50 years) will undergo urine sample pregnancy testing prior to X-ray imaging. A pilot study with 20 participants will be conducted first. Experiences from the pilot will be used to refine the study protocol if needed. If modifications are made, they will be subjected to ethics review and will be provided on ClinicalTrials.gov. After the pilot study, the researchers aim to recruit an additional 80 patients (totaling up to 100 participants).

Our research questions are 1) What is the prevalence of radiologically confirmed needle retention among PWIDs*? The secondary research questions are

1. Do patient-reported symptoms and the suspicion of a retained needle fragments correspond to radiologically confirmed needle retention?
2. What are the predisposing factors to needle fragmentation?
3. Have PWIDs sought medical attention prior to the study for possible symptoms in the injection sites?
4. How frequently are verified needle fragments surgically removed within five years after their detection, and are verified needle fragments a proxy or a risk factor for mortality? *As only patients in outpatient care will be recruited, the sample is not entirely representative of all PWIDs in the study area (e.g., people who are hospitalized or imprisoned are not recruited).

ELIGIBILITY:
Inclusion Criteria:

* History of intravenous drug use
* Current treatment of the drug abuse problem at a local low-threshold drug abuse service unit or primary health care centre.
* Adherence to fill in the questionnaire
* Participation to X-ray imaging of injection sites

Exclusion Criteria:

* No history of intravenous drug use
* Does not adhere to fill in the questionnaire or refuses X-ray imaging
* Pregnancy
* Underage (18 years old)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population base is the adult IVD users from the drug abuse treatment centres in Tampere, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of needle fragment retentions among intravenous drug users. | An average of 2 years.
  The prevalence of needle fragment retentions among intravenous drug users. The number of individuals with at least one radiologically confirmed needle fragment in subcutaneous tissue over the total number of participants.
Risk factors for needle fragment retentions in a cross-sectional design | An average of 2 years.
  Risk factors for needle fragment retentions in a cross-sectional design. Patient characteristics as risk factors for having subcutaneous needle fragment retentions.
The proportion of patients with surgically removed needle fragment retentions at five years of follow-up. | Up to 5 years.
  The proportion of patients with surgically removed needle fragment retentions after five years of follow-up. Patients with needle fragment retentions will be referred to the surgical clinic and will be prospectively followed up through healthcare records.

CONTACTS AND LOCATIONS:
Overall Officials: Otso Arponen, MD-PhD, Study Chair — Pirkanmaa Hospital District (PSHP); Olli PO Nevalainen, MD-PhD, Study Chair — City of Tampere; Tampere University; Pirkanmaa Hospital District (PSHP).; Irina Rinta-Kiikka, MD-PhD, Study Chair — Tampere University Hospital; Heidi Laukkala, MD, Study Chair — City of Tampere, Tampere University; Markku Sumanen, MD-PhD, Principal Investigator — Tampere University
Locations (1):
- Hatanpää Health Center, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No
No plans to share individual-level data with other investigators.

REFERENCES:
- [Derived] Laukkala H, Arponen O, Rinta-Kiikka I, Sumanen M, Nevalainen OPO. Prevalence and predisposing factors of retained drug needle fragments in people who inject drugs: a protocol for a preliminary cross-sectional multicentre observational study in Finland. BMJ Open. 2025 Aug 10;15(8):e099521. doi: 10.1136/bmjopen-2025-099521. PMID 40784774